CLINICAL TRIAL: NCT03003975
Title: Efficacy of Single Versus Double Cryoballoon Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation (SD-Cryo-AF): A Randomized Study
Brief Title: Single Versus Double Cryoballoon Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation
Acronym: SD-CRYO-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Carina Blomstrom Lundqvist, Professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SD-CRYO-AF
Record Dates: First submitted 2016-12-09; First posted 2016-12-28 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Cryoballoon; Achieve
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI by single cryoballoon application (Active Comparator): A single cryoballoon application for pulmonary vein isolation will be guided by a Multipolar Recording Catheter (Achieve Mapping Catheter), passed through the inner lumen of the cryoablation catheter. A single application of 4 minutes will be used per vein guided by recording of loss of electrograms and by a defined drop of temperature within 2 minutes application. If a stable position with adequate occlusion of the vein the Achieve catheter should be located proximally for evaluation of entrance block during application, but can be advanced deeper for stability and then retracted to the ostium to evaluate vein isolation (entrance block).
  If the vein then is isolated after a single application, the operator can move on to the next vein.
  Interventions: Device: PVI by single cryoballoon application guided by Achieve Mapping Catheter
- PVI by 2 cryo applications (Active Comparator): Cryoballoon ablation with a conventional guidewire passed through the inner lumen of the catheter for stability will be used. Ablation will be performed with 2 consecutive applications for 4 minutes each in each vein guided by degree of occlusion and temperature drop at the discretion of the physician.
  Interventions: Device: PVI by 2 routine cryoballoon applications

INTERVENTIONS:
Device: PVI by single cryoballoon application guided by Achieve Mapping Catheter — Pulmonary vein isolation by single cryoballoon application guided by recorded electrogram signals from an internal Mapping Catheter and by temperature drop if mapping of signals is not possible (temperature cutoff < or = -40 degrees C)
  Other Names: Arctic Front™ Advance Cardiac CryoAblation Catheter; Achieve Mapping Catheter
  Arms: PVI by single cryoballoon application
Device: PVI by 2 routine cryoballoon applications — Pulmonary vein isolation by 2 cryoballoon applications guided by degree of occlusion and by temperature drop according to discretion of physician
  Other Names: Arctic Front™ Advance Cardiac CryoAblation Catheter
  Arms: PVI by 2 cryo applications

SUMMARY:
This is a clinical study where the investigators will assess the efficacy of a single cryoballoon application per vein guided by a multipolar recording catheter as compared with a conventional technique with 2 cryoballoon applications for pulmonary vein isolation (PVI) in patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
This is a prospective, randomized clinical study performed at one centre. The objective is to assess the efficacy of a single cryoballoon application per vein guided by a multipolar recording catheter as compared with a conventional technique with 2 cryoballoon applications for pulmonary vein isolation in patients with atrial fibrillation (AF).

140 subjects with paroxysmal or persistent atrial fibrillation referred for their first AF ablation procedures will be enrolled.

Recruitment, ablation and follow-up will be performed at Dep of Cardiology in Uppsala University Hospital, Uppsala, Sweden.

Study duration is 2 years with 12--months enrolment period and 1 year follow-up per subject.

Pulmonary vein isolation (PVI) will be performed using the Arctic Front Advance cryoballoon ablation catheter. Patients will be randomized to a single cryoballoon application guided by a multipolar recording catheter or to a conventional technique with 2 cryoballoon applications. After cryoballoon ablation of all pulmonary veins, PV conduction block will be assessed by a separate circular mapping catheter. Acute procedural success is defined as complete electrical isolation of a pulmonary vein assessed by entrance and exit block, including 20 minutes waiting time. Complications and duration of the procedure will be assessed.

Patients will be followed at three, six and 12 months after the ablation procedure. A 12 lead ECG, a 7 day Holter monitoring, quality of life (EQ5D) and EHRA score, will be performed at baseline, 6 and 12 months. as well as Biomarkers including nTproBNP and troponin I, will be performed at baseline, and at 6 and 12 months (only nTproBNP). Predictive variables for successful outcome/AF recurrence will be analysed.

The frequency of symptomatic recurrence of AF and number of reablations will be compared at 6 and 12 months, and in those requiring a redo ablation procedure the status of PV reconduction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent AF verified by ECG
* Patients with symptoms corresponding to at least Europe Heart Rhythm Association (EHRA) score 2.

Exclusion Criteria:

* Sinus rhythm cannot be maintained for at least one hour after an electrical cardioversion.
* Congestive heart failure with New York Heart Association (NYHA) class 3 or more.
* Left ventricular ejection fraction < 35% not secondary to AF with inadequate rate control, according to the judgement of the investigator.
* Left atrial diameter ≥ 55 mm judged by transthoracic echocardiography.
* Prior AF ablation procedure.
* Longstanding persistent AF
* AF secondary to a transient or correctable abnormality including electrolyte imbalance, trauma, recent surgery, infection, toxic ingestion, and uncontrolled thyroid disease as well as AF triggered by other uniform supraventricular tachycardia.
* Contraindication to treatment with anticoagulants.
* Significant valvular disease or planned cardiac intervention.
* Hypertrophic cardiomyopathy.
* Recent cardiac disease states within the last 6 months; unstable angina, acute myocardial infarction, revascularisation procedures, valve disease
* Implantable cardioverter-defibrillator (ICD), cardiac resynchronization therapy (CRT) device.
* Dual chamber- and single chamber-pacemaker when the patient is pacemaker dependent on ventricular level
* Patients with contraindications for transseptal catheterization or appropriate vascular access is precluded.
* Renal failure requiring dialysis or abnormalities of liver function tests.
* Participant in investigational clinical or device trial.
* Unwilling or unable to give informed consent or inaccessible for follow-up and psychological problem that might limit compliance.
* Active abuse of alcohol or other substance which may be causative of AF and/or might affect compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Frequency of acute pulmonary vein isolation after first ablation. | Acute during ablation procedure
  Frequency of complete pulmonary vein isolation after first pass of ablation as per protocol

SECONDARY OUTCOMES:
Procedure time | During ablation procedure
  Procedure time of AF ablation (from initial puncture to removal of sheaths)
Fluoroscopy exposure | During ablation procedure
  Total time of fluoroscopy for AF ablation
Freedom from atrial fibrillation | Evaluated after 12 months
  No atrial fibrillation after first ablation
Adverse/Serious Adverse events | Evaluated after 12 months
  Complications during and after ablation
Quality of Life after ablation | Evaluated after 12 months
  Quality of life assessed by EQ5D after ablation compared to baseline
Reduction of symptom severity score after ablation | Evaluated after 12 months
  Symptoms Severity Questionnaire, score reduction after ablation
Reduction of overall symptoms of atrial fibrillation after ablation | Evaluated after 12 months
  Symptom assessed by EHRA Symptom Classification score reduction after ablation
Cost of ablation procedure | Evaluated after initial ablation (within 24 h after ablation)
  Assessed by time for procedure, used resources and equipment during/after ablation
Quality of life after ablation (measured as EQ5D score) | Evaluated after 12 months
  EQ5D measured before ablation and after 12 months
Hospitalisation after ablation | Evaluated after 12 months
  hospitalisation (no of days)
Maximum troponin I (ng/L) levels after ablation as a predictor of clinical success | Evaluated after 12 months
  Maximum troponin I (ng/L) levels as a predictor of freedom from AF after 12 months
Nt-proBNP levels before ablation as a predictor of clinical success | Evaluated after 12 months
  Nt-proBNP levels as a predictor of freedom from AF after 12 months
Left atrial diameter (mm) before ablation as a predictor of clinical success | Evaluated after 12 months
  Left atrial diameter in mm (LAX view) as a predictor of freedom from AF after 12 months
Left atrial volume (ml/m2) before ablation as a predictor of clinical success | Evaluated after 12 months
  Left atrial volume (ml/m2) as a predictor of freedom from AF after 12 months
Age (years) as a predictor of clinical success | Evaluated after 12 months
  Age at ablation (years) as a predictor of freedom from AF after 12 months; 2 groups; < 70 and >70 years old
Sex as a predictor of clinical success | Evaluated after 12 months
  Sex as a predictor of freedom from AF after 12 months. 2 groups; male vs females
CHADsVASc score as a predictor of clinical success | Evaluated after 12 months
  CHADsVASc score as a predictor of freedom from AF after 12 months
BMI (kg/m2) as a predictor of clinical success | Evaluated after 12 months
  BMI (kg/m2) as a predictor of freedom from AF after 12 months
Atrial conduction time as a predictor of clinical success | Evaluated after 12 months
  Mean conduction time over left atrium as a predictor of freedom from AF after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carina Blomström Lundqvist, Professor, Principal Investigator — Uppsala University
Locations (1):
- Department of Cardiology, University Hospital in Uppsala, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No